CLINICAL TRIAL: NCT06454487
Title: Investigating the Effectiveness and Acceptability of Isometric Handgrip Training in Remote Cardiac Rehabilitation Patients: A Randomized Controlled Trial With an Embedded Qualitative Study
Brief Title: Exploring IHG Training in CR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Windsor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReDA13269
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cardiac Rehabilitation; Blood Pressure
Keywords: Cardiac Rehabilitation; Hand Grip Training; Blood Pressure
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CR+IHG (Experimental): Cardiac Rehabilitation (usual care) PLUS Isometric Hand grip training
  Interventions: Other: Isometric Hand Grip Training
- CR (Active Comparator): Cardiac Rehabilitation (usual care) Only
  Interventions: Other: CR

INTERVENTIONS:
Other: Isometric Hand Grip Training — IHG training will be performed with an inflatable ball three days per week for 12 weeks (with at least a day of rest between each session) with intensity set based on RPE (Borg CR-10 scale).
  Other Names: IHG
  Arms: CR+IHG
Other: CR — Standard of Care
  Other Names: Cardiac Rehabilitation
  Arms: CR

SUMMARY:
Research has shown that isometric (constant squeeze) exercise training using an isometric handgrip (IHG) device lowers resting blood pressure (BP) in those with and without high BP. The purpose of this study is to explore if IHG training will lower resting BP in people doing cardiac rehabilitation more than doing only cardiac rehabilitation. Once eligibility is confirmed participants will be randomly assigned to one of two groups for the study. One group will do IHG training in addition to cardiac rehabilitation (Group 1), and the other group will do only cardiac rehabilitation (Group 2). Participants assigned to Group 1 will be asked to do IHG training on their own with an inflatable ball three days per week for 12 weeks with intensity set based on rating of perceived exertion (RPE) or rating of effort. Participants will self-measure and report their resting BP to investigators. The acceptability of doing IHG training will also be explored by conducting interviews with participants as will the impact that IHG training may have on psychological wellbeing by administering surveys to participants.

ELIGIBILITY:
Inclusion Criteria:

* Component adult (greater ≥ 18 years) who can provide informed consent.
* Proficient in English (speaking, writing, and reading).
* Medically cleared by the cardiac rehabilitation program to participate in exercise-based cardiac rehabilitation.
* History of only coronary artery disease, the most common cardiovascular disease (CVD), which may include individuals with a previous myocardial infarction and/or procedure such as a percutaneous coronary intervention and/or coronary artery bypass grafting.
* Minimum of "blue" level of technology capability (assigned by the cardiac rehabilitation program) indicating ability to use a phone and email for correspondence. Note: The majority of individuals who enroll in the cardiac rehabilitation program are assigned to this level.
* No physical limitation(s) that would hinder the performance of isometric handgrip training.
* Access to a blood pressure monitoring device to record at home measures.

Exclusion Criteria:

* If the participant does not meet the inclusion criteria (identified above).
* Moreover if an individual has a history of a CVD or disease-related complications (e.g., heart failure, atrial fibrillation, ventricular arrhythmias, aortic aneurysm, valve repair and/or replacement) and/or related procedures (e.g., placement of a pacemaker and/or implantable cardiac defibrillator) that is not coronary artery disease (as described in the inclusion criteria) they will be excluded.

Note: Individuals may have other comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Resting Blood Pressure | 12 weeks
  Self report of Resting Blood Pressure at baseline vs week 5, 9 and post-intervention

SECONDARY OUTCOMES:
User Experience of IHG | 12 weeks
  Qualitative content analysis (participant interviews)
Psychological state | 12 weeks
  Self-report of depression, anxiety, stress, and mindfulness using participant surveys

CONTACTS AND LOCATIONS:
Overall Officials: Cheri McGowan, PhD, Principal Investigator — Windsor University and LawsonHRI
Locations (2):
- Canada (2):
  - St Joseph's Hospital Cardiac Rehabilitation and Secondary Prevention, London, Ontario
  - Hotel Dieu Grace Cardiac Rehabilitation, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD